CLINICAL TRIAL: NCT04367337
Title: Health Behavior Change During COVID-19 Pandemic: the Focus on Handwashing
Brief Title: Health Behavior Change During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: 3228-1BPSYPSBEH-30
Record Dates: First submitted 2020-04-28; First posted 2020-04-29 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2020-08

CONDITIONS: Health Behavior
Keywords: General population; Adult; Handwashing; Social cognition; Anxiety; COVID-19
MeSH Terms: conditions — Health Behavior; Anxiety Disorders; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (14):
- Poland: Adults, general population, N = 400
  Interventions: Other: No intervention
- Australia: Adults, general population, N = 400
  Interventions: Other: No intervention
- Canada: Adults, general population, N = 400
  Interventions: Other: No intervention
- China: Adults, general population, N = 400
  Interventions: Other: No intervention
- France: Adults, general population, N = 400
  Interventions: Other: No intervention
- Gambia: Adults, general population, N = 400
  Interventions: Other: No intervention
- Germany: Adults, general population, N = 400
  Interventions: Other: No intervention
- Israel: Adults, general population, N = 400
  Interventions: Other: No intervention
- Italy: Adults, general population, N = 400
  Interventions: Other: No intervention
- Malaysia: Adults, general population, N = 400
  Interventions: Other: No intervention
- Portugal: Adults, general population, N = 400
  Interventions: Other: No intervention
- Romania: Adults, general population, N = 400
  Interventions: Other: No intervention
- Singapore: Adults, general population, N = 400
  Interventions: Other: No intervention
- Switzerland: Adults, general population, N = 400
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational data collection only, accounting for COVID-19 morbidity and mortality levels within each country

SUMMARY:
This study aims at investigating handwashing behavior during COVID-19 pandemic. It was hypothesized that social-cognitive and emotional predictors as well as COVID-19 morbidity and mortality rates within the country would be associated with handwashing behavior in the general population of adults in 14 countries.

DETAILED DESCRIPTION:
This observational study aims at testing the adherence to handwashing guidelines (the World Health Organization, WHO, 2020) at two measurement points, spanning 1 month. Adults from the general population in 14 countries (Poland, Australia, Canada, China, France, Gambia, Germany, Israel, Italy, Malaysia, Portugal, Romania, Singapore, Switzerland) will provide self-report data on handwashing behavior and its social-cognitive predictors (perceived effectiveness of handwashing, risk perception, outcome expectancy, self-efficacy, intention, planning, and action control), anxiety, as well as COVID-19 morbidity and mortality rates within the country.

ELIGIBILITY:
Inclusion Criteria:

* adults (from general population) who provided informed consent to participate

Exclusion Criteria:

* younger than <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults in 14 countries are recruited using the snowballing method. Data are collected using an online platform (software: Qualtricts).
Sampling Method: Non-Probability Sample
Enrollment: 6079 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Handwashing adherence | 1 month
  The 12-item self-report measure of adherence to handwashing guidelines across situations (e.g., after visiting public spaces, after touching garbage, etc.) based on the guidelines issued by the World Health Organization and the Centers for Disease Control and Prevention. The responses are provided on a 4-point scale, ranging from 1 (strongly disagree) to 4 (strongly agree). Higher scores indicate better outcomes (the higher level of adherence to handwashing guidelines).
Frequency of handwashing | 1 month
  The 1-item self-report measure of the frequency of handwashing (for at least 20 seconds, all surfaces of the hands) daily. The responses are provided on a 4-point scale, ranging from 1 (less than once) to 5 (more than 10 times). Higher scores indicate better outcomes (the higher frequency of handwashing).

SECONDARY OUTCOMES:
Self-efficacy | 1 month
  4 self-efficacy questionnaire items; mean item score ranging from 1 to 4, higher scores indicate stronger self-efficacy
Risk perception | 1 month
  3 questionnaire items to assess risk perception; mean item score ranging from 1 to 5, higher scores indicate higher risk perception
Outcome expectancy | 1 month
  4 items assessing positive (1 item) and negative (1 items) outcome expectancies; mean item scores ranging from 1 to 4, higher scores indicate more positive outcome expectancies
Intention | 1 month
  2 questionnaire items assessing intention to adhere to handwashing recommendations; mean item scores ranging from 1 to 4, higher scores indicate stronger intention to wash hands (for at least 20 seconds, all surfaces of the hands)
Planning | 1 month
  2 questionnaire items assessing action planning (1 item) and coping planning (1 item); mean item scores ranging from 1 to 4, higher scores indicate a higher level of self-reported planning
Action control | 1 month
  3 questionnaire items assessing a facet of action control, namely self-monitoring; mean item scores ranging from 1 to 4, higher scores indicate a higher level of self-reported monitoring of handwashing behavior
Perceived effectiveness of hand hygiene | 1 month
  1 questionnaire item assessing perceptions of handwashing as an effective means of preventing coronavirus SARS-CoV-2 infection; item scores ranging from 1 to 4, higher scores indicate a higher level of perceived effectiveness of hand hygiene
Anxiety | 1 month
  7-item self-report scale (Generalized Anxiety Disorder, GAD-7) scale to assess anxiety symptoms; mean item scores ranging from 1 to 4, higher scores indicate a higher level of generalized anxiety
Country-level COVID-19 morbidity and mortality rates | 60 days
  The daily cumulative numbers for COVID-19 morbidity and mortality in the study countries. Published daily as the Situation Report by World Health Organization, starting on 21 January 2020. Higher numbers indicate the higher cumulative COVID-19 morbidity and mortality rates in the country.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Luszczynska, PhD, Principal Investigator — SWPS University of Social Sciences and Humanities
Locations (14):
- the University of Melbourne, Melbourne, Australia
- University of New Brunswick, Fredericton, Canada
- Peking University, Beijing, China
- University of Bordeaux, Bordeaux, France
- Freie Universität Berlin, Berlin, Germany
- Bar-Ilan University, Ramat Gan, Israel
- University of Padova, Padua, Italy
- Perdana University, Serdang, Malaysia
- SWPS University of Social Sciences and Humanities, Wroclaw, Lower Silezia, Poland
- University of Lisbon, Lisbon, Portugal
- Babes-Bolyai Unversity, Cluj-Napoca, Romania
- Nanyang Technological University, Singapore, Singapore
- University of Zurich, Zurich, Switzerland
- London School of Hygiene and Tropical Medicine (in collaboration with MRC Unit The Gambia at LSHTM), Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: Undecided
The lead researchers in 14 countries will have full access to data collected across the countries.
  In line with the Consortium Agreement (v2, 16th Jul 2020) data will be openly available under following conditions:
  De-identified individual participant data that underline the results reported in publications; individual-level aggregated data (e.g., sum scores for scales) used for main analyses in respective publications; available following the publication, no end date of availability; available for analyses that are conducted to achieve aims in the approved proposal.
  Due to local regulations, there are exceptions in terms of data sharing rules (stated above):
  * AUSTRALIA: Data from Australia will be available for 5 years after collection.
  * GERMANY, SWITZERLAND: Instead of individual-level sum scores, variance-covariance matrices will be shared.
  * MALAYSIA: Data will not be shared.

REFERENCES:
- [Background] World Health Organization. Coronavirus disease (COVID-19) advice for the public. 2020. https://www.who.int/emergencies/diseases/novel-coronavirus-2019/advice-for-public
- [Background] Centers for Disease Control and Prevention. When and how to wash your hands. 2020. https://www.cdc.gov/handwashing/when-how-handwashing.html
- [Background] Reyes Fernandez B, Knoll N, Hamilton K, Schwarzer R. Social-cognitive antecedents of hand washing: Action control bridges the planning-behaviour gap. Psychol Health. 2016 Aug;31(8):993-1004. doi: 10.1080/08870446.2016.1174236. Epub 2016 Apr 26. PMID 27049339
- [Background] Schwarzer R, Lippke S, Luszczynska A. Mechanisms of health behavior change in persons with chronic illness or disability: the Health Action Process Approach (HAPA). Rehabil Psychol. 2011 Aug;56(3):161-70. doi: 10.1037/a0024509. PMID 21767036
- [Background] Ruiter RAC, Abraham C, Kok G. Scary warnings and rational precautions: A review of the psychology of fear appeals. Psychol Health. 2011;11(1): 613-630. doi: 10.1080/08870440108405863
- [Derived] Szczuka Z, Siwa M, Abraham C, Baban A, Brooks S, Cipolletta S, Danso E, Dombrowski SU, Gan Y, Gaspar T, Gaspar de Matos M, Griva K, Jongenelis M, Keller J, Knoll N, Ma J, Abdul Awal Miah M, Morgan K, Peraud W, Quintard B, Shah V, Schenkel K, Scholz U, Schwarzer R, Taut D, Tomaino SCM, Vilchinsky N, Wolf H, Luszczynska A. Handwashing adherence during the COVID-19 pandemic: A longitudinal study based on protection motivation theory. Soc Sci Med. 2023 Jan;317:115569. doi: 10.1016/j.socscimed.2022.115569. Epub 2022 Nov 21. PMID 36436259
- [Derived] Luszczynska A, Szczuka Z, Abraham C, Baban A, Brooks S, Cipolletta S, Danso E, Dombrowski SU, Gan Y, Gaspar T, de Matos MG, Griva K, Jongenelis MI, Keller J, Knoll N, Ma J, Miah MAA, Morgan K, Peraud W, Quintard B, Shah V, Schenkel K, Scholz U, Schwarzer R, Siwa M, Taut D, Tomaino SCM, Vilchinsky N, Wolf H. The Interplay Between Strictness of Policies and Individuals' Self-Regulatory Efforts: Associations with Handwashing During the COVID-19 Pandemic. Ann Behav Med. 2022 Apr 2;56(4):368-380. doi: 10.1093/abm/kaab102. PMID 34871341
- [Derived] Szczuka Z, Abraham C, Baban A, Brooks S, Cipolletta S, Danso E, Dombrowski SU, Gan Y, Gaspar T, de Matos MG, Griva K, Jongenelis M, Keller J, Knoll N, Ma J, Miah MAA, Morgan K, Peraud W, Quintard B, Shah V, Schenkel K, Scholz U, Schwarzer R, Siwa M, Szymanski K, Taut D, Tomaino SCM, Vilchinsky N, Wolf H, Luszczynska A. The trajectory of COVID-19 pandemic and handwashing adherence: findings from 14 countries. BMC Public Health. 2021 Oct 5;21(1):1791. doi: 10.1186/s12889-021-11822-5. PMID 34610808